CLINICAL TRIAL: NCT01604473
Title: Endothelial Function and Arterio-Venous Fistula Maturation
Acronym: EFAVF
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-02538
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; CKD; ESRD; AV Fistula; Arterio-venous fistula; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease: Individuals with Chronic Kidney Disease stages IV or V anticipating the need for hemodialysis access through an arterio-venous fistula.

SUMMARY:
An arterio-venous fistula is a surgical procedure that supports access for people undergoing hemodialysis (HD) for End Stage Renal Disease (ESRD). This observational pilot study seeks to better understand the factors that contribute to the successful maturation of an arterio-venous fistula. A primary aim of this study is to see if endothelial function (the biochemical events initiated by cells lining the arteries) is associated with successful maturation. Other aims include determining if pro-inflammatory markers in the blood or evidence of gene expression are associated with successful maturation.

DETAILED DESCRIPTION:
Current practice guidelines stipulate that 65% of all prevalent ESRD patients should receive HD through some sort of arterio-venous fistula (AVF). An AVF is a subcutaneous, permanent vascular access created surgically by connecting a vein with an artery and is the preferred mode of access due to lower rates of infection or thrombosis compared to prosthetic grafts or tunneled lines. An AVF is mature if it can sustain high quality HD. However, rates of primary failure (the inability of an AVF to sustain HD) are high, ranging from 40-70%. Traditional coronary risk factors such as hypertension, hypercholesterolemia, and diabetes mellitus, have limited ability to allow surgeons to predict which AVFs will mature.

One possible explanation involves vascular remodeling, the structural changes which occur in a blood vessel in response to hemodynamic stimuli. The endothelial, lying at the interface of the vessel wall and flowing blood, is a "biosensor", responding to changes in blood flow and pressure. It initiates a complex biological response including cellular proliferation and migration, matrix degradation, and cellular apoptosis. This longitudinal, observational study hypothesizes that endothelial function is a critical modulator of AVF maturation. Specifically, that patients with inflammation will have impaired endothelial function and demonstrate less significant remodeling than others.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease classification Stage IV or V
* Adequate quality cephalic or basilic vein based on pre-operative assessment
* Able to provide written informed consent
* Able to travel to the SFVA Medical Center or UCSF Medical Center for follow-up examination

Exclusion Criteria:

* Age >90 or < 18 years
* Diagnosed hypercoaguble state
* Recent surgery or other major illness or infection within 6 weeks
* Use of immunosuppresive medication
* History or organ transplantation
* Pregnancy or plans to become pregnant
* Estimated life expectancy is less than 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04-29 (Actual); Study Completion 2014-04-29 (Actual)

PRIMARY OUTCOMES:
Maturation of Arteriovenous Fistula | 90 days
  Maturation is defined by either:
  * Less than three months have elapsed since AVF creation and cannulation of the fistual with two 17 gauge needles and delivery of a minimum of 400 ml/min for the duration of dialysis
  * Greater than three months have elapsed since AVF creation and the individual has not yet initiated hemodialysis and the vein diameter is 4 mm and the volumetric flow rate is 400 ml/min.

SECONDARY OUTCOMES:
Primary Patency | 90 days
  Primary patency of the AV fistula
Secondary Patency | 90 days
  Secondary patency of the AV fistula
Stenosis of AV fistula | 90 days
  Moderate or severe stenosos of AV fistual as detected by duplex ultrasound or fistulagram
Venous remodeling | 90 days
  Venous remodeling at 3 months
Arterial remodeling | 90 days
  Arterial remodeling at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Warren J Gasper, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco Medical Center, San Francisco, California